CLINICAL TRIAL: NCT07120230
Title: Evaluation of the Safety and Rapid Recovery Effect of the Tubeless Strategy in Lung Transplantation: A Prospective Single-Arm Clinical Study
Brief Title: Tubeless Strategy in Lung Transplantation: A Prospective Single-Arm Study
Acronym: Tubeless-LTx-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Dean, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tubeless-LTx-2025; Tubeless-LTx-2025 (Registry Identifier: Evaluation of the safety and rapid recovery effect of the tubeless strategy in lung transplantation)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lung Transplant Recipient

STUDY DESIGN:
Masking Description: Outcomes were assessed using predefined criteria; where feasible, assessors performing outcome adjudication were not involved in perioperative airway management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tubeless LTx Group (Experimental): Participants in this group will receive lung transplantation surgery without standard tracheal intubation. Instead, they will breathe on their own using a special airway device called a laryngeal mask airway (LMA), combined with a bronchial blocker to separate lung ventilation during surgery. Sedation is maintained with intravenous medications (propofol, remifentanil, and dexmedetomidine), and participants will remain spontaneously breathing or receive minimal breathing assistance as needed. The surgical incision will be numbed using local anesthesia with lidocaine and ropivacaine injections. After surgery, the LMA will be removed in the operating room, and participants will transition directly to non-invasive breathing support before being monitored in the ICU.
  Interventions: Procedure: Tubeless Lung Transplantation Surgery

INTERVENTIONS:
Procedure: Tubeless Lung Transplantation Surgery — Patients undergoing this surgery receive lung transplantation surgery without standard tracheal intubation. Instead, they will breathe on their own using a special airway device called a laryngeal mask airway (LMA), combined with a bronchial blocker to separate lung ventilation during surgery. Sedation is maintained with intravenous medications (propofol, remifentanil, and dexmedetomidine), and participants will remain spontaneously breathing or receive minimal breathing assistance as needed. The surgical incision will be numbed using local anesthesia with lidocaine and ropivacaine injections. After surgery, the LMA will be removed in the operating room, and participants will transition directly to non-invasive breathing support before being monitored in the ICU.

SUMMARY:
This prospective, single-center, single-arm study evaluates the feasibility, safety, and rapid recovery outcomes of a tubeless strategy in lung transplantation. Consecutive eligible adult lung transplant recipients undergo lung transplantation without standard endotracheal intubation, using a laryngeal mask airway and standardized regional anesthesia and intravenous sedation protocols.

The primary outcome is freedom from invasive ventilation in the operating room, defined as removal of the airway device before leaving the operating room with no reinstitution of invasive ventilation within 72 hours. Secondary outcomes include postoperative ICU length of stay, postoperative hospital length of stay, postoperative invasive ventilation requirement, postoperative complications (assessed up to 30 days), and perioperative mortality.

DETAILED DESCRIPTION:
The study was initially registered as a randomized controlled trial. However, randomization was not feasible due to patient refusal of treatment allocation. Therefore, the study proceeded as a prospective single-arm cohort with consecutive enrollment. Outcome definitions remained unchanged. The study was conducted at a single center.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily participate in this study, possess full civil capacity, be able to understand the study protocol, and sign a written informed consent.
2. Be between 18 and 74 years of age.
3. Be listed on the lung transplant waiting list of the China Lung Transplant Registry (CLuTR) or their respective centers and intend to undergo lung transplantation.
4. Have an American Society of Anesthesiologists (ASA) anesthesia grade 4 or lower and be expected to be able to tolerate anesthesia.
5. Preoperative assessment indicates that cardiac function (LVEF ≥ 50%), renal function (eGFR ≥ 60 mL/min/1.73 m²), and liver function (Child-Pugh A) are compatible with surgery. 6) Completed the pre-lung transplant respiratory rehabilitation program assessment and demonstrated good compliance;

7) Not receiving continuous endotracheal intubation or venovenous extracorporeal membrane oxygenation (ECMO) support prior to surgery; 8) No active infection, including active tuberculosis, HIV, or positive hepatitis B/C viral load before surgery; 9) Have a clear and reliable post-operative care support system (including at least one primary caregiver).

Exclusion Criteria:

1. Refusing to sign informed consent or withdrawing informed consent during the trial;
2. Planning to undergo a second lung transplant or a combined multi-organ transplant (such as heart-lung, lung-liver, lung-kidney, etc.);
3. Clearly combined with uncontrollable active infection (such as tuberculosis, uncontrolled fungal infection) or sepsis;
4. Patients with obvious neuropsychiatric disorders, unconsciousness or long-term use of sedative/analgesic psychotropic drugs before surgery;
5. Active malignant tumors (except those treated within the past 2 years) or those with a high risk of postoperative recurrence;
6. Clearly diagnosed severe chest deformity or spinal deformity that may affect lung compliance during surgery;
7. Serum anti-HLA high sensitization (PRA ≥ 80%) and no matching donor available;
8. There are clear contraindications to the planned tubeless surgical anesthesia strategy (such as expected intraoperative airway difficulty, pharyngeal stenosis and laryngeal mask unsuitable, etc.);
9. BMI ≥ 30 kg/m² or < 16 kg/m². 10) Pregnant or lactating women.

11) Other conditions deemed unsuitable for participation in this study by the investigator (e.g., anticipated inability to complete follow-up, concurrent malignancy, etc.).

12) Patients with bronchiectasis or bronchial vascular hyperplasia difficult to manage with interventional therapy prior to surgery.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Freedom from invasive ventilation in the operating room | From end of surgery (postoperative day 0) through 72 hours postoperatively (up to 72 hours).
  Proportion of participants who have the airway device removed before leaving the operating room and do not require reinstitution of invasive ventilation within 72 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No